CLINICAL TRIAL: NCT01328834
Title: Efficacy and Safety of Tacrolimus Sustained-release Capsules in Induction Treatment in Refractory Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Xueqing Yu, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGLN-003
Record Dates: First submitted 2011-02-01; First posted 2011-04-05 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-10

CONDITIONS: Nephritis, Lupus
Keywords: Nephritis, Lupus; Tacrolimus
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVAGRAF (Experimental): Tacrolimus Sustained-release Capsules (ADVAGRAF) treatment in induction phase
  Interventions: Drug: Tacrolimus Sustained-release Capsules (ADVAGRAF)

INTERVENTIONS:
Drug: Tacrolimus Sustained-release Capsules (ADVAGRAF) — Started: 0.05-0.1mg/kg/d, one time per day, the blood level 5-10ng/ml in the induction treatment.
  Other Names: ADVAGRAF: Tacrolimus Sustained-release Capsules

SUMMARY:
This a pilot study to evaluate the efficacy and safety of Tacrolimus Sustained-release Capsules (ADVAGRAF) treatment for the induction therapy of refractory lupus nephritis (LN).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, 14-65 years of age;
2. Diagnosis of SLE according to the ACR criteria (1997);
3. Kidney biopsy within the 6 months prior to study with a histologic diagnosis (ISN/RPS 2003 classification of LN) class IV, V, V+ III, V+ IV;
4. Usage of intravenous pulse cyclophosphamide for more than 3 times or immunosuppression therapy (AZA, MMF, oral cyclophosphamide, ect) for more than 6 months;
5. proteinuria > 1g/24hr or Scr > 1.3 mg/dl or active urinary sediment (erythrocyte cast, > 5 WBC/high power field (hpf) (excluding infection), > 5 RBC/hpf);
6. Provision of written informed consent by subject or guardian

Exclusion Criteria:

1. Inability or unwillingness to provide written informed consent ;
2. Usage of immunosuppression therapy (MMF, CTX, CysA, MTX etc) for more than 1 week within 1 month or intravenous MP Pulse treatment prior to entry;
3. Scr > 4mg/dl (354umol/L);
4. Needing pulse intravenous MP or intravenous immunoglobulin;
5. Lupus encephalopathy;
6. Diagnosed DM; Malignant tumors (except fully cured basal cell carcinoma);
7. History of significant gastrointestinal disorders (e.g. active peptic ulcer disease or pancreatitis) within 3 month prior to enter this study;
8. Known hypersensitivity or contraindication to tacrolimus, corticosteroids
9. Any Active systemic infection or history of serious infection within one month of entry or known infection with HIV, hepatitis B, or hepatitis C;
10. Participation in another clinic trial and/or receipt of investigational drugs within 4 weeks prior to screening;
11. Pregnancy, nursing or use of a non-reliable method of contraception.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Remission rate (complete or partial remission) | 6 months after therapy

SECONDARY OUTCOMES:
The changes of proteinuria | every 3 months up to 6 months
SLEDAI scores | every 3 months up to 6 months
  SLEDAI:Systemic Lupus Erythematosus Disease Activity Index (Bombardier et al, 1992).
Number of participants with adverse events as a measure of safety and tolerability | every 3 months up to 6 months
  Adverse events, including infections, transient increases in serum creatinine, gastrointestinal complaints, liver function disorder and glucose intolerance, etc.
The changes of renal function | every 3 months up to 6 months
Relapse | every 3 months up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xueqing, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University IRB, Guangzhou, Guangdong, China